CLINICAL TRIAL: NCT01760772
Title: The Role of GLP-1 in Lipid Metabolism in Healthy Subjects and in Subjects After Bariatric Surgery
Brief Title: Effect of GLP-1 on Postprandial Lipid Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: David Dalessio (Other)
Responsible Party: Sponsor-Investigator, David Dalessio, Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-09-20-01
Record Dates: First submitted 2012-11-17; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-11

CONDITIONS: Heart Disease
Keywords: heart disease; GLP-1; Exendin-9; postprandial lipids
MeSH Terms: conditions — Heart Diseases | interventions — exendin (9-39); Injections; Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator): 0.9% saline
  Interventions: Other: saline
- Exendin-9 (Ex-9) (Experimental): Bolus of Ex-9 (7,500 pmol/kg) followed by a continuous infusion at 750 pmol/kg/min
  Interventions: Drug: Exendin-9
- GLP-1 (Experimental): GLP-1 infusion at 0.3 pmol/kg/min
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: Exendin-9 — Bolus of Ex-9 (7500 pmol/kg) over 1 minute followed by continuous infusion at 750 pmol/kg/min
  Other Names: Synthetic exendin (9-39) injection
  Arms: Exendin-9 (Ex-9)
Drug: GLP-1 — Constant infusion of GLP-1 at 0.3 pmol/kg/min
  Other Names: 7-36 amide
  Arms: GLP-1
Other: saline — Constant infusion
  Arms: Saline

SUMMARY:
Individuals with obesity have an increased risk for heart disease and diabetes. There are current drugs on the market that target the hormone, Glucagon like peptide-1 (GLP-1) to treat diabetes. The investigators want to determine if targeting this hormone will also help people with high cholesterol and triglycerides. In this study, the investigators are looking at the role of GLP-1 in healthy subjects and subjects that have had bariatric surgery.

DETAILED DESCRIPTION:
Major consequences of the global pandemic of obesity include cardiovascular disease, type 2 diabetes and dyslipidemia. The dyslipidemia of obesity commonly consists of fasting hypertriglyceridemia with increased plasma very low-density lipoprotein (VLDL), reduced high-density lipoprotein (HDL) and the presence of small, dense low-density lipoprotein (LDL). However, more recently, increased secretion of intestinally derived lipoproteins (LPs) has been recognized as contributing to this dyslipidemic profile and postprandial lipemia has been linked to adverse health outcomes. Glucagon-like peptide-1 (GLP-1), a hormone secreted during meal absorption that plays a key role in the control of plasma glucose has been implicated as a candidate hormone for regulating intestinal lipid metabolism. Studies in rodents demonstrate that treatment with the GLP-1R agonist; exendin-4 (Ex-4) reduced postprandial chylomicron (CM) production and CM-associated cholesterol and triglyceride (TG). Similar results were found in Type 2 diabetes (T2D) subjects treated with Ex-4; in these reports there was a reduction in both intestinally derived LP production and total plasma TG. The objective of this study is to determine whether GLP-1 is involved in the physiologic regulation of postprandial lipid metabolism in healthy women, and to test the hypothesis that the improved lipid parameters found in overweight women who have had bariatric surgery are mediated by GLP-1. The specific aims for this project will 1) determine if either pharmacologic treatment with GLP-1 and/or antagonism of endogenous GLP-1 activity improves postprandial lipid metabolism in healthy subjects and 2) determine the role of elevated postprandial GLP-1 levels on lipid metabolism in obese subjects who have had a sleeve gastrectomy. The investigators will use infusions of synthetic GLP-1 with the native hormone to confirm the lipid-lowering results that have been published using pharmacologic GLP-1 receptor (GLP-1R) agonists. The investigators will also use the GLP-1R antagonist exendin-(9-39) to determine the role of endogenous GLP-1 on lipemia after a test meal. A demonstration that this is a physiologic action would expand the current understanding of lipid metabolism, provide new insight into the effects of bariatric surgery, and allow the design of more refined, mechanistic studies of this process. In addition, the potential for GLP-1R signaling to promote lipid metabolism has direct translational importance in that therapies already exist that could capitalize on this mechanism. Understanding the role of GLP-1R regulation of lipid absorption and clearance could lead to more appropriate targeting of GLP-1 based drugs to specific diabetic patients, i.e. ones with problematic dyslipidemia and higher risk for cardiovascular disease. Moreover, understanding the effects of GLP-1 on plasma lipids could eventually lead to new approaches for treating nondiabetic dyslipidemic persons.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: Healthy, normolipemic men and postmenopausal women; aged 40-60 years; BMI between 25-35
* Aim 2: Men and postmenopausal women after successful vertical sleeve gastrectomy (VSG) surgery and age- and weight-matched non-surgical control men and postmenopausal women; ages between 40-6- years; BMI between 28-35; steady weight for at least 3 months prior to study

Exclusion Criteria:

Exclusion Criteria for Aim 1:

* History or clinical evidence of impaired fasting glucose or diabetes mellitus, myocardial infarction or symptoms of congestive heart failure, history or active liver or renal disease, calculated glomerular filtration rate < 60 mL/min).
* History of extreme dyslipidemia (i.e. familial hypercholesterolemia) or Cardiovascular disease (CVD).
* Fasting plasma total cholesterol > 200 mg/dL and fasting plasma TGs > 150 mg/dL.
* Surgery within 6 months.
* Pregnancy or lactation.
* Anemia defined as hematocrit < 33%.
* History of cancer or anorexia nervosa or GI disorders.
* Use of medications that alter insulin sensitivity (i.e. niacin, glucocorticoids, metformin) or lipid metabolism (i.e. statin, niacin, fibrate, ezetimibe).
* Plasma HbA1c > 6.0.
* Fasting glucose > 110 mg/dL
* Electrocardiogram (ECG) abnormalities: evidence of ischemia or arrhythmia.

Exclusion Criteria for Aim 2:

* History of CVD.
* Fasting plasma total cholesterol > 250 mg/dL and fasting plasma TGs > 300 mg/dL.
* Surgical intervention within 6 months.
* Anemia defined as hematocrit < 33%.
* History of cancer or anorexia nervosa or other major GI disease or surgery.
* Use of medications that alter insulin sensitivity (i.e. niacin, glucocorticoids, metformin) or lipid metabolism (i.e. statin, ezetimibe).
* HbA1c > 6.0.
* Fasting glucose > 110 mg/dL
* Electrocardiogram (ECG) abnormalities: evidence of ischemia or arrhythmia.
* Significant renal, hepatic or pulmonary disease.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Postprandial Lipids Levels and Apolipoprotein B (ApoB) Levels in plasma | 2 years
  Total and lipoprotein-associated triglyceride and cholesterol levels in baseline and postprandial plasma.
  Total apolipoprotein B48 (ApoB48) and apolipoprotein B100 (ApoB100) levels in baseline and postprandial plasma.

SECONDARY OUTCOMES:
Plasma insulin and glucagon | 2 years
  Plasma insulin and glucagon in the fasting and postprandial periods
Plasma free fatty acid (FFA) and glucose levels | 2 years
  Plasma FFA and glucose levels during the fasting and postprandial state
Plasma d-xylose and acetaminophen levels | 2 years
  Plasma d-xylose and acetaminophen levels as indices of gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Adams, PhD, Principal Investigator — University of Cincinnati; David D'Alessio, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Veteran's Affairs Clinical Research Unit, Cincinnati, Ohio, United States